CLINICAL TRIAL: NCT05596799
Title: Facing Eating Disorder Fears for Anorexia Nervosa: a Virtual Relapse Prevention Program Targeted At Approach and Avoidance Behaviors
Brief Title: Facing Eating Disorder Fears for Anorexia Nervosa
Acronym: FED-F
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Cheri Levinson, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#: 21.0992; 1R34MH126965-01A1 (NIH)
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Eating Disorders; Anorexia Nervosa; Anorexia Nervosa in Remission
Keywords: therapy; eating disorder; anorexia nervosa; treatment; relapse prevention; virtual treatment
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Facing Eating Disorder Fears Condition (Experimental): Participants will complete 1 session of education about the treatment. After completion of treatment education and baseline questionnaires, participants will complete sessions 2 through 12 of virtual treatment for anorexia nervosa and mobile assessments.
  Interventions: Behavioral: Facing Eating Disorder Fears Condition
- Treatment as Usual (No Intervention): Participants will complete baseline measures, mobile assessments and treatment as usual.

INTERVENTIONS:
Behavioral: Facing Eating Disorder Fears Condition — The first session consists of diagnosis and general psychoeducation on anorexia nervosa and treatment for anorexia nervosa. After psychoeducation and baseline questionnaires are complete, sessions 2-12 include exposure-based virtual treatment for common eating disorder fears (food, weight gain, body sensations, and social situations).
  Arms: Facing Eating Disorder Fears Condition

SUMMARY:
FED-F is a modular treatment that enhances exposure therapy with psychoeducation and cognitive skills teaching how to face fears of (a) food, (b) weight gain, (c) interoception/body, and (d) social situations. The study goals are to (1) refine and test the acceptability and feasibility of FED-F treatment (Phase I), (2) test if this treatment outperforms treatment as usual (TAU) delivered post-acute treatment as adjunctive to stepdown specialty care (Phase II), and (3) to examine if treatment targets the hypothesized mechanism of action: approach behaviors (Phase II). These goals will lead to a highly deployable and accessible virtual treatment targeted at core AN mechanisms that predict relapse. Specific aims are to (1) refine FED-F into a fully virtual format with input from patients and stakeholders and collect preliminary data (N=10) on its feasibility and acceptability (Phase I), (2) conduct a small pilot RCT (randomized controlled trial) of FED-F (n=30) as compared to TAU (n=30; Phase II), and (3) examine if FED-F targets approach/avoidance behaviors and test if this mechanism is associated with clinical outcomes (Phase II).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Meets criteria for DSM-5 defined AN, AN partial remission, or AN full remission, Atypical Anorexia Nervosa (AAN), AAN partial remission, or AAN full remission
* Has been discharged from intensive (i.e., inpatient, residential, or partial hospital program) in the past 6 months

Exclusion Criteria:

* Under 18
* Over 65
* Does not meet criteria for DSM-5 defined AN, AN partial-remission, or AN full-remission
* High and active Suicidality
* Active Mania
* Active psychosis
* Medically Compromised Status including extremely low weight (less than or equal to 75% median BMI for age, sex, and height)
* Does not meet criteria for DSM-5 defined AN, AN partial remission, or AN full remission, AAN, AAN partial remission, or AAN full remission
* Has not been discharged from intensive (i.e., inpatient, residential, or partial hospital program) in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Structured Clinical Interview for DSM-5 (SCID-5) | Up to 2-month follow-up
  The SCID-5 is a semi-structured interview used to arrive at DSM-5 diagnoses. Participants will complete the ED, anxiety, depression, mania, psychosis, and suicide modules. SCID-5 has strong psychometric properties.
Change in Eating Disorder Fear Inventory (EFI) | Up to 2-month follow-up
  EFI is a semi-structured interview used to assess ED fears, such as fear of weight gain, food, and associated consequences. It will be used to generate fears to focus on during treatment and comprehensively assesses all domains of ED fear.
Change in Treatment Interview | Up to 2-month follow-up
  The Treatment Interview will assess all current and past treatment experiences (partial hospitalization, residential, etc.), as well as dates of treatment. It will also assess primary type of treatment (CBT vs supportive), as well as current usage of psychotropic medications and duration of illness.
Change in Eating Disorder Examination Questionnaire 6.0 (EDE-Q) | Up to 2-month follow-up
  The EDE-Q assesses ED behaviors, thoughts, and outcomes (e.g., fasting, binge eating). The EDE-Q has demonstrated excellent test-retest reliability, internal consistency, good criterion validity and concurrent validity.
Change in Fear of Food Measure (FOFM) | Up to 2-month follow-up
  The FOFM is a measure that assesses three cognitive-behavioral dimensions of fear of food: anxiety about food, food avoidance behaviors, and feared concerns (e.g., fear of weight gain). It has strong factor, convergent, divergent, and construct validity.
Change in Eating Disorder Fear Questionnaire (EFQ) | Up to 2-month follow-up
  The EFQ is a measure of five central ED fears: fear of weight gain, fear of social eating, fear of physical sensations, fear of social consequences (from gaining weight), fear of personal consequences (from gaining weight). EFQ has strong factor, convergent, and construct validity and assesses multiple domains of ED fear.

SECONDARY OUTCOMES:
Change in Behavioral Approach Task | Up to 2-month follow-up
  The Behavioral Approach Task will be used at each diagnostic assessment. It is a standardized behavioral rating task adapted from Ritzert (2017) for use with specific phobias. This task asks participants to rate their anxiety and likelihood to avoid feared stimuli (e.g., pizza, grocery stores, tight jeans) and is adapted from behavioral ratings obtained when building an exposure hierarchy for the treatment of AN fear, which has been implemented in over 200 patients with AN.
Change in Behavioral Inhibition System/Behavioral Activation System (BIS/BAS) | Up to 2-month follow-up
  The Behavioral Inhibition System/Behavioral Activation System will assess avoidance and approach tendencies with a well-validated and established measure.
Change in Subjective Units of Distress (SUDS) | Up to session 12
  SUDS is a behavioral measure used during exposure treatment to measure anxiety and will be collected throughout each treatment session. The SUDS scale has been shown to be a valid and reliable measure of state anxiety. SUDS ratings can range from 0 (completely calm) to 100 (highest anxiety).
Change in State Fear of Food Measure | Up to Session 12
  The state version of the fear of food measure, which assesses food anxiety, food avoidance, and feared concerns (e.g., weight gain), will be used during sessions. This measure will be collected at the beginning and end of each therapy session.
Change in Mobile Assessment of Approach and Avoidance | Up to Session 12
  Real-world approach and avoidance behaviors will be assessed via mobile assessment. While momentary assessment is a newer and more innovative method of assessing approach tendencies, the usage of self-report, behavioral, and momentary data will provide the opportunity to compare assessment methodologies in preparation for usage in a larger R01 RCT.

CONTACTS AND LOCATIONS:
Overall Officials: Cheri A Levinson, Ph.D., Principal Investigator — University of Louisville
Locations (1):
- Eating Anxiety Laboratory and Clinic, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews G, Cuijpers P, Craske MG, McEvoy P, Titov N. Computer therapy for the anxiety and depressive disorders is effective, acceptable and practical health care: a meta-analysis. PLoS One. 2010 Oct 13;5(10):e13196. doi: 10.1371/journal.pone.0013196. PMID 20967242
- [Background] Carl JR, Miller CB, Henry AL, Davis ML, Stott R, Smits JAJ, Emsley R, Gu J, Shin O, Otto MW, Craske MG, Saunders KEA, Goodwin GM, Espie CA. Efficacy of digital cognitive behavioral therapy for moderate-to-severe symptoms of generalized anxiety disorder: A randomized controlled trial. Depress Anxiety. 2020 Dec;37(12):1168-1178. doi: 10.1002/da.23079. Epub 2020 Jul 29. PMID 32725848
- [Background] Levinson CA, Christian C, Ram SS, Vanzhula I, Brosof LC, Michelson LP, Williams BM. Eating disorder symptoms and core eating disorder fears decrease during online imaginal exposure therapy for eating disorders. J Affect Disord. 2020 Nov 1;276:585-591. doi: 10.1016/j.jad.2020.07.075. Epub 2020 Jul 21. PMID 32794449
- [Background] Farrell NR, Brosof LC, Vanzhula IA, Christian C, Bowie OR, Levinson CA. [Exploring Mechanisms of Action in Exposure-Based Cognitive Behavioral Therapy for Eating Disorders: The Role of Eating-Related Fears and Body-Related Safety Behaviors]. Behav Ther. 2019 Nov;50(6):1125-1135. doi: 10.1016/j.beth.2019.01.008. Epub 2019 Feb 12. French. PMID 31735247
- [Background] Butler RM, Heimberg RG. Exposure therapy for eating disorders: A systematic review. Clin Psychol Rev. 2020 Jun;78:101851. doi: 10.1016/j.cpr.2020.101851. Epub 2020 Mar 21. PMID 32224363